## **Informed Consent Form**

The Role of Probiotics L. Plantarum, S. thermophiles, B. bifidum on Gut Inflammation, Bacterial Translocation, and CD4+ Cell Count in HIV Patients with Immunological Non-Responder (PIONIR)



## **INVESTIGATORS:**

Principal : Erni Juwita Nelwan, MD, Ph.D

Others: Rina Agustina, MD, M.Sc., Ph.D

Prof. Marcellus Simadibrata, MD, Ph.D

**FACULTY OF MEDICINE** 

**Universitas Indonesia** 

Approved October 30th, 2017



**RSUPN Dr. Cipto Mangunkusumo**Jl. Diponegoro No. 71 Jakarta 10430
Telp: (021) 3918301 Fax: (021) 3148991

MRN Name Sex Date of Birth

(Please fill in the blank or put the ID sticker here)

| Principal Investigator : Erni J. Nelwan, MD, Ph.D Informant : Subject Name : Date of Birth (Age) : Sex Address : | INFORMED CONSENT FORM |
|---|---|
| Subject Name : Date of Birth (Age) : Sex : | |
| Name : Date of Birth (Age) : Sex : | |
| Date of Birth (Age) : : : | |
| Sex : | |
| Δddroee | |
| Phone Number (Cellphone) | |
| | RK |
| 1 Title of The Study The Role of Probiotics Lactobacillus | |
| plantarum, Streptococcus thermophiles, Bifidobacterium bifidum on Gut | |
| Inflammation, Bacterial Translocation, and | |
| CD4+ Cell Count in HIV Patients with | |
| Immunological Non-Responder: Double | |
| Blind Randomized Controlled Trial | |
| 2 Objectives of The Study To determine the effects of probiotics (good | |
| bacteria) Lactobacillus plantarum, | |
| Streptococcus thermophilus dan | |
| Bifidobacterium bifidum in HIV patients with | |
| immune response failure | |
| 3 Methods of The Study You will be asked about HIV disease, | |
| physically examined, fill HIV symptoms | |
| index form, and have your blood tested for | |
| immune cells (CD4+ and Th17) level, viral | |
| load level, and bacteria translocation marker | |
| (16SrRNA) level. You will also have your | |
| stool tested for gut inflammation marker | |
| (fecal calprotectin) level and gut cells | |
| (colonocytes) level. | |
| We will take 12 cc of blood for test sample. | |
| You will get candies which you need to | |
| chew, 1 (one) tablet each day for 12 | |
| (twelve) weeks. ARV medication should be | |
| continued as usual, but should not be taken | |
| with the candies in the same time in a day. | |
| You will be examined physically and have | |



**RSUPN Dr. Cipto Mangunkusumo**Jl. Diponegoro No. 71 Jakarta 10430
Telp: (021) 3918301 Fax: (021) 3148991

MRN Name Sex Date of Birth

(Please fill in the blank or put the ID sticker here)

| | | the same laboratory tests as in the beginning of the study. This is a voluntary study. You may not |
|---|---|---|
| | | participate in this study and it will not affect |
| | | your treatment in Cipto Mangunkusumo |
| | | National Central General Hospital. |
| 4 | Total of Subject | 80 people |
| 5 | Time of Study | 1 (one) year with 12 weeks intervention |
| 6 | Significances of Study | This study will bear the cost of laboratory |
| | (Including to Study | study including CD4+, viral load, Th17, |
| | Subjects) | 16SrRNA levels by blood test and fecal |
| | | calprotectin and colonocytes levels by fecal |
| | | test. These tests will be conducted 2 (two) |
| | | times. This study will help doctors in understanding |
| | | HIV patients with immune response failure |
| | | thus increasing the quality of practice. |
| 7 | Risks and Adverse Events | The risk is pain at area of blood sampling. |
| | of The Study | The adverse events that may occur |
| | · | including nausea, vomiting, diarrhea which |
| | | may cause lack of body fluid, and |
| | | lactobacilemia which may cause fever and |
| | | severe stomachache. |
| 8 | Study Subject | You need to consume the candies with the |
| | Inconvenience | flavor you do not like every day for 12 |
| 0 | Adverse Event | (twelve) weeks. |
| 9 | Compensation | If there is any lactobacilemia symptom, sepsis protocol will be executed and the |
| | Compensation | probiotics treatment will be stopped. |
| | | If there is lack of body fluid, a procedure of |
| | | fluid therapy will be executed and probiotics |
| | | treatment will be stopped. |
| 10 | Alternative Managements | You may not participate in this study and |
| | (if occurred) | take the ARV treatment as usual. |



MRN : Name : Sex : Date of Birth :

(Please fill in the blank or put the ID sticker here)

| | TYPE OF INFORMATION | CONTENT OF INFORMATION | MARK |
|---|---|---|---|
| 11 | Data Confidentiality | All your information will be kept and will not | |
| | | be given to any unauthorized person related | |
| | | to your treatment. | |
| 12 | Cost to Subjects | No cost will be borne by subjects | |
| 13 | Incentive for Subjects | No incentive will be given to subjects | |
| 14 | Name, Address, and<br>Phone Number of Principal<br>Investigator | Erni J. Nelwan, MD, Ph.D<br>Divisi Penyakit Tropik dan Infeksi,<br>Departemen Ilmu Penyakit Dalam, FKUI-<br>RSCM<br>Cellphone no: 021-3914190; 0811961229 | |

I have received information in page 1, 2, and 3 about the study conducted by Erni J. Nelwan, MD, Ph.D titled The Role of Probiotics *Lactobacillus plantarum, Streptococcus thermophiles, Bifidobacterium bifidum* on Gut Inflammation, Bacterial Translocation, and CD4+ Cell Count in HIV Patients with Immunological Non-Responder: Double Blind Randomized Controlled Trial. I clearly understand the information.

By signing this form, I agree to participate in the study voluntarily without any threat from anyone. I have right to cancel this agreement if I feel being harmed in any way.

| Subject's Signature or Thumbprint | Date |
|--------------------------------------|------|
| Subject's Name | |
| Subject's Guardian/Witness Signature | Date |

Subject's Guardian/Witness Name

Note: Subject's Guardian/Witness Signature is needed if the subject is illiterate, having a decreased consciousness, having mental disorder, or under 18 years old.



MRN :
Name :
Sex :
Date of Birth :
(Please fill in the blank or put the ID sticker here)

| I have given the information to | subject appropriate | ely and truthfully | about the stud | dy obje | ctives, |
|---|---|---|---|---|---|
| significances, procedure, and | potential risk and | uncomforting si | ituation which | may h | appen |
| (detailed information provided). | I also have answer | red the question | ns related to the | e study | in the |
| best possible way. | | | | | |
| Investigator's Signature | | Date | | | |
| Investigator's Name | | | | | |